CLINICAL TRIAL: NCT01783223
Title: Prevalence of Chronic Inebriates to the Emergency Department and Suitability for Sobering House Services
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 12-3560
Record Dates: First submitted 2013-01-23; First posted 2013-02-04 (Estimated); Results first posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intoxicated patients: patients in the Emergency Department who appear to be intoxicated with ethanol.

SUMMARY:
This study is intended to evaluate the prevalence of chronically inebriated patients in the Emergeny Department (ED). Patients will be identified prospectively by screening all patients (24/7) presenting to the ED for one month. A running tally of all patients in the ED will be kept. Of these patients, any patient that is noted to have alcohol intoxication will be identified. The chart of that patient will be reviewed for details about the patient's alcohol use and for the patient's suitability for a sobering house, which is a place where intoxicated patients can go to await sobriety. The chart will also be reviewed for the number of previous visits for alcohol use to our hospital ever and in the last year.

DETAILED DESCRIPTION:
For this cross-sectional study, all patients presenting to the ED of an urban, Level 1 trauma center for one month were prospectively screened by trained research associates. When an intoxicated patient was identified, study information including patient demographics, diagnoses, vital signs, blood alcohol concentration (BAC), GCS on arrival, ability to ambulate independently on arrival, use of physical or chemical restraint, previous ED visits, length of stay, and health insurance was collected. Data was analyzed using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the emergency department for alcohol intoxication

Exclusion Criteria:

* Under 18
* Prisoners
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the emergency department for alcohol intoxication
Sampling Method: Non-Probability Sample
Enrollment: 668 (Actual)
Dates: Start 2012-11; Primary Completion 2018-06-26 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Miner, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intoxicated Patients
Started | 668
Completed | 668
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intoxicated Patients
Number analyzed (Participants) | 668
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 588
  >=65 years | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [33 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264
  Male | 404
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Intoxicated Patients Eligible for a Sobering House
Description: Determine the proportion of patients in the emergency department that are intoxicated and how many of those would be eligible to go to a sobering house. Eligibility for a sobering house is at the discretion of the treating physician and includes the ability to ambulate without assistance and no further acute need for medical treatments.
Time Frame: Eligibility for a sobering house is assessed during the current ED admission. The study ends when patient is discharged from the ED, an expected average time of 9 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Intoxicated Patients
Number analyzed (Participants) | 668
Participants | 163

ADVERSE EVENTS:
Time Frame: 1824 minutes
Arm/Group | Intoxicated Patients
All-Cause Mortality (participants affected / at risk) | 0/668
Serious Adverse Events (participants affected / at risk) | 50/668
Other Adverse Events (participants affected / at risk) | 505/668
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intoxicated Patients (N=668)
hospital admission (Nervous system disorders) | 44 (44) — admitted to the hospital for care related to alcohol intoxication during emergency department observation period
endotracheal intubation (Respiratory, thoracic and mediastinal disorders) | 6 (6) — intubation during observation in emergency department
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intoxicated Patients (N=668)
unable to ambulate independently or provide basic medical information (Nervous system disorders) | 180 (180) — during ED observation period
agitation requiring physical restraint (Nervous system disorders) | 276 (276) — during ED observation
agitation requiring sedation (Nervous system disorders) | 283 (283) — during ED observation period
procedure performed (Surgical and medical procedures) | 122 (122) — during ED observation period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2011-03-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT01783223/Prot_000.pdf